CLINICAL TRIAL: NCT06528587
Title: Rehabilitation of Single Aesthetic Areas Using Narrow Diameter Implants With Computer Guided Implant Insertion: a Prospective Study
Brief Title: Rehabilitation of Single Aesthetic Areas Using Narrow Diameter Implants
Acronym: IDR
Status: Completed | Type: Observational
Sponsor: Fondazione Policlinico Universitario Agostino Gemelli IRCCS (Other)
Responsible Party: Sponsor
Other Study IDs: 6683
Record Dates: First submitted 2024-07-08; First posted 2024-07-30 (Actual); Last update posted 2026-01-08 (Actual); Status verified 2024-07

CONDITIONS: Implant Complication
Keywords: narrow diameter implant

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- narrow diameter implant: Patients who have performed computer-guided implant surgery for the rehabilitation of single edentulism in the anterior region with lack of adequate bone thickness or mesio-distal space using implants with narrow diameter.
  Interventions: Procedure: narrow diameter implant

INTERVENTIONS:
Procedure: narrow diameter implant — Rehabilitation of single edentulism in the anterior region with narrow diameter implants and computer guided surgery.

SUMMARY:
The scientific literature does not provide scientific evidence on how to manage patients suffering from monoedentulism with ridges having a reduced bone thickness or a reduced mesio-distal space. Narrow diameter implants could be a solution to rehabilitate patients suffering from these clinical conditions while avoiding longer, more complex and sometimes even multidisciplinary therapies. However, there is a lack of clinical studies analyzing the outcomes of rehabilitation with narrow diameter implants.

DETAILED DESCRIPTION:
Dental implants are considered a predictable rehabilitation option in the event of tooth extraction or missing tooth. In some cases, the inevitable resorption of the alveolar ridge after tooth extraction can make the insertion of dental implants difficult or even impossible without the use of more advanced bone regeneration procedures. Narrow diameter implants represent an alternative treatment option in areas with limited ridge width. Narrow alveolar ridges and limited interdental or inter-implant spaces continue to pose a challenge to the clinician. In the case of a narrow ridge, two options are available: the first option is to insert a standard diameter implant following bone augmentation procedures; the second option is to use an implant with a narrow diameter. Regarding the mesio-distal gap, an adequate distance between teeth and implants is necessary to reduce subsequent bone resorption and recession of the papillae. Difficult clinical situations with limited mesio-distal space or reduced ridge width can be overcome by using narrow diameter implants. Correct three-dimensional implant positioning is the key factor to obtain, in addition to good integration, favorable prosthetic results and a good long-term aesthetic result. To optimize the insertion of the implants, reducing the intrinsic imprecision of the conventional free-hand technique, computer-guided static surgery protocols can be used to plan the angulation, position and depth of the implant with a digital software. Narrow diameter implants therefore have their own indication for the replacement of lateral incisors of the maxilla and for the incisors of the mandible.

ELIGIBILITY:
Inclusion Criteria:

* Patients who have undergone implant surgery to perform implant rehabilitation of single edentulism in the anterior region to insert a reduced diameter implant;

  * ASA I and ASA II patients;
  * Age > 18yr;
  * Non-smokers or smokers ≤ 5 cig/day;
  * Achievement of FMPS and FMBS ≤ 15%;
  * Signing of the written informed consent to participate in the study.

Exclusion Criteria:

* Severe general medical pathologies;

  * Immunodeficiency states;
  * Radiotherapy in the head and neck region;
  * Uncontrolled diabetes or hypertension;
  * Smokers >5 cigs/day;
  * Impossibility to carry out homogeneous and continuous follow-up;
  * Documented allergy to the biomaterials used;
  * Pregnancy or breastfeeding;
  * Inability to provide written informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients aged >18 years, in good general health, who have undergone implant rehabilitation of single edentulism in the anterior region will be selected.
Sampling Method: Non-Probability Sample
Enrollment: 17 (Actual)
Dates: Start 2024-09-01 (Actual); Primary Completion 2025-11-01 (Actual); Study Completion 2025-11-01 (Actual)

PRIMARY OUTCOMES:
peri-implant marginal bone loss in millimeters | 12 months from implant placement
  evaluation of the peri-implant marginal bone loss in millimeters

SECONDARY OUTCOMES:
soft tissue evaluation in millimeters | 12 months from implant placement
  evaluation of marginal soft tissues levels in millimeters
biological complication rate in percentage | 12 months from implant placement
  evaluation of biological complications in percentage
esthetics | 12 months from implant placement
  evaluation of the esthetics using the PES score
mechanical complication rate in percentage | 12 months from implant placement
  evaluation of mechanical complications in percentage

CONTACTS AND LOCATIONS:
Overall Officials: Paolo Francesco Manicone, Principal Investigator — Fondazione Policlinico Universitario A. Gemelli, IRCCS
Locations (1):
- Fondazione Policlinico Universitario A. Gemelli IRCCS, Rome, Roma, Italy

IPD SHARING:
Plan to Share IPD: No